CLINICAL TRIAL: NCT03356015
Title: Comparison of the Efficacy and Tolerability Between 3-L and 4-L Polyethylene Glycol in Bowel Preparation
Brief Title: Comparison Between 3-L and 4-L Polyethylene Glycol in Bowel Preparation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Director of Gastroenterology Dept and Digestive Endoscopy Center, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: PEG-171116
Record Dates: First submitted 2017-11-20; First posted 2017-11-29 (Actual); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Bowel Preparation Scale; Adenoma Detection Rate
Keywords: Polyp detection rate; Adenoma detection rate; Boston Bowel Preparation Scale
MeSH Terms: interventions — Polyethylene Glycols

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4L Polyethylene Glycol (Experimental): 4L-group received 4 bags of PEG and were instructed to drink 2L at 19:00 in the evening before the day of colonoscopy at a rate of 250 mL every 15 minutes, and to drink the remaining 2L 4 to 6 h before colonoscopy at the same rate.
  Interventions: Drug: 4L Polyethylene Glycol
- 3L Polyethylene Glycol (Active Comparator): 3L-group received 3 bags of PEG and were instructed to drink 1L at 19:00 in the evening before the day of colonoscopy at a rate of 250 mL every 15 minutes, and to drink the remaining 2L 4 to 6 h before colonoscopy at the same rate.
  Interventions: Drug: 3L Polyethylene Glycol

INTERVENTIONS:
Drug: 4L Polyethylene Glycol — 4L group received double-dose PEG at 19:00 in the evening before the day of colonoscopy at a rate of 250 mL every 15 minutes.
  Arms: 4L Polyethylene Glycol
Drug: 3L Polyethylene Glycol — 3L group were instructed to drink 1L PEG at 19:00 in the evening before the day of colonoscopy at a rate of 250 mL every 15 minutes
  Arms: 3L Polyethylene Glycol

SUMMARY:
High quality bowel preparation is essential for successful colonoscopy. This study aimed to assess the impact of the dose of Polyethylene Glycol(PEG) on the quality of bowel preparation. This prospective, endoscopist-blinded, randomized, controlled study was conducted. 3L-group received 3 bags of PEG and were instructed to drink 1L at 19:00 in the evening before the day of colonoscopy at a rate of 250 mL every 15 minutes, and to drink the remaining 2L 4 to 6 h before colonoscopy at the same rate. 4L-group received 4bags of PEG and were instructed to drink 2 L at 19:00 in the evening before the day of colonoscopy at a rate of 250 mL every 15 minutes, and to drink the remaining 2L 4 to 6 h before colonoscopy at the same rate. The primary outcome was the quality of the bowel preparation according to the Boston Bowel Preparation Scale (BBPS). The secondary outcomes included polyp detection rate (PDR), adenoma detection rate (ADR), tolerance, and subjective feelings of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients aged 18-75 years
2. Referred for routine diagnostic colonoscopy
3. Patients who have signed inform consent form

Exclusion Criteria:

1. pregnancy or breastfeeding
2. allergy to purgatives
3. suspected intestinal obstruction, stricture, or perforation
4. hemodynamic instability
5. impaired swallowing reflex or mental status
6. severely medical status, such as New York Heart Association grade III or grade IV congestive heart failure and severe renal failure
7. history of oesophagus、stomach 、duodenum、small intestine or colorectal surgery
8. participation declined.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2018-01-01 (Estimated); Study Completion 2018-02-01 (Estimated)

PRIMARY OUTCOMES:
the Boston Bowel Preparation Scale | 2 days
  The primary end point of the study was adequate bowel preparation quality de ned as a BBPS total score of ≥6 with all segment scores ≥2

SECONDARY OUTCOMES:
Polyp detection rate | 2 days
  The secondary end point of the study included polyp detection rate
Adenoma detection rate | 2 days
  The secondary end point of the study included adenoma detection rate
The mean number of incremental adenomas | 2 days
  It was a new metric called ADR-Plus, the mean number of incremental adenomas after the fist.

CONTACTS AND LOCATIONS:
Overall Officials: Peng Cheng, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Second Military Medical University, Shanghai, China

REFERENCES:
- [Derived] Cheng P, Chen Q, Li J, Pang L, Feng C, Wang N, Bai Y, Li Z, Meng X. 3 liters of polyethylene glycol vs. standard bowel preparation have equal efficacy in a Chinese population: a randomized, controlled trial. Am J Transl Res. 2022 Aug 15;14(8):5641-5650. eCollection 2022. PMID 36105041